CLINICAL TRIAL: NCT03819868
Title: Efficacy of Resin Sealing in Deciduous and Permanent Molars: Split-mouth Randomized Clinical Trial
Brief Title: Efficacy of Sealing Molars: Split-mouth Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD, Senior Lecturer, Clinical Professor, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLM 5
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Dental Caries
Keywords: dental caries; molars; Pit and Fissure Sealants
MeSH Terms: conditions — Dental Caries; Van der Woude syndrome | interventions — Technology, High-Cost

STUDY DESIGN:
Intervention Model Description: Split-mouth
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Cost (Active Comparator): Restoration using a high-cost sealant
  Interventions: Procedure: High cost
- Low Cost (Experimental): Restoration using a low-cost sealant
  Interventions: Procedure: Low Cost

INTERVENTIONS:
Procedure: High cost — Surfaces allocated to this group will be treated with a high-cost sealant (Fluroshield®, Dentsply, São Paulo, Brazil), according to the manufacturer's instructions.
  Arms: High Cost
Procedure: Low Cost — Surfaces allocated to this group will be treated with a low-cost sealant (Prevent®, FGM Produtos Odontológicos, Santa Catarina, Brazil), according to the manufacturer's instructions.
  Arms: Low Cost

SUMMARY:
The sealing of fossae and fissures is an effective procedure in preventing occlusal caries lesions. However, there are gaps regarding its efficacy in the treatment of initial enamel lesions. In addition, there are no studies in the literature that have compared the longevity of sealings performed with the different sealants available in the market. Thus, the objective of this study is to evaluate the efficacy of fossae and fissures sealings performed with a low-cost resinous sealant in occlusal lesions in enamel in permanent and deciduous molars. This is a multicenter clinical study of non-inferiority, randomized, controlled, double blind (patient and operator) with 60 deciduous molars and 340 permanent molars of children 4 and 9 years of age. The sample unit will be the tooth, which will be randomized into two groups using a distributed randomization list in mixed envelopes that will be open only at the time of the procedure. The teeth allocated in the test group will be treated with the sealant preventâ; Those allocated in the control group will employ the Fluroshieldâ sealant. In both groups the procedure will follow the manufacturer's standards. The efficacy of the sealant will be evaluated by means of clinical and radiographic control at 6, 12 and 18 months after the procedure. Secondary outcomes, such as retention, cost, acceptability and quality of life, will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least two deciduous and/or permanent molars with occlusal caries lesions scores 1, 2 or 3 of the Icdas (Ismail et al., 2007) will be included, one on each side, preferably from the same arch.

Exclusion Criteria:

* Patients with special needs;
* using orthodontic appliances;
* with systemic diseases;
* Teeth that present restorations, sealants, formation defects, deep caries lesions that may lead to pulp impairment;
* teeth with fistula and/or abscess;
* teeth with spontaneous painful symptomatology.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dental caries progression | Every 6 months up to 18 months
  Caries progression will be evaluated radiographically by three previously trained evaluators (through theoretical classes and evaluation of 13 clinical photographs) and calibrated. These examiners will not know the chronological order and compare the images two to two first by two evaluators and when there is disagreement between the two, the third examiner shall be called for tie-breaker. The possible progression of the treated caries lesion will be codified as:
  * Present progression: Increased radiolucidity area of the Lesion
  * Absent progression: No increase in the area of radiolucidity of the lesion.

SECONDARY OUTCOMES:
Cost-effectiveness | 18 months
  The costs of each treatment procedure will be calculated and compared with thresholds values for intervention costeffectiveness by region, determined by World Health Organization (http://www.who.int/choice/costs/CER_levels/en/).
Impact on children's quality of life | Baseline and 18 months
  The oral health related quality of life will be measured using a validated questionnaire according to the children's age. The "Early Childhood Oral Health Impact Scale" (ECOHIS) (Tesch et al., 2008) will be applied with 4-5 years old children. The "Child Perceptions Questionnaire" (CPQ) will be used for 6-9 years old children (Martins et al., 2009).
  They will be applied immediately before the procedure and on 18 months follow-up and we will measure the difference between answers at baseline and the end of treatment (18months)
Children self-reported discomfort | Baseline
  The discomfort of each treatment will be evaluated using the facial scale of Wong-Baker (Wong, Baker, 1988). The patient will be asked to choose the face that is more similar to how he/she felt during the treatment. The answer should be given solely by the child, which means no parental or professional interferences. Each face corresponds to a number, within a numeric scale from 0 to 5, with 0 no discomfort and 5 the greatest discomfort. At the end, the averages of each score will be compared between the experimental groups.
Sealant retention | Every 6 months up to 18 months
  The elements submitted to the treatment will be codified in accordance with Hesse et al. (2012):
  * Full retention: When the restorer material was Intact when subjected to clinical examination;
  * Partial loss: When there was a loss of a part of the restorer material previously applied;
  * Total Loss: When the restorer material has been lost in its entirety.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Sao Leopoldo Mandic, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hesse D, Bonifacio CC, Mendes FM, Braga MM, Imparato JC, Raggio DP. Sealing versus partial caries removal in primary molars: a randomized clinical trial. BMC Oral Health. 2014 May 28;14:58. doi: 10.1186/1472-6831-14-58. PMID 24884684
- [Result] Martins MT, Ferreira FM, Oliveira AC, Paiva SM, Vale MP, Allison PJ, Pordeus IA. Preliminary validation of the Brazilian version of the Child Perceptions Questionnaire 8-10. Eur J Paediatr Dent. 2009 Sep;10(3):135-40. PMID 19761288
- [Result] Tesch FC, Oliveira BH, Leao A. [Semantic equivalence of the Brazilian version of the Early Childhood Oral Health Impact Scale]. Cad Saude Publica. 2008 Aug;24(8):1897-909. doi: 10.1590/s0102-311x2008000800018. Portuguese. PMID 18709230
- [Result] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Result] Pitts N, Melo P, Martignon S, Ekstrand K, Ismail A. Caries risk assessment, diagnosis and synthesis in the context of a European Core Curriculum in Cariology. Eur J Dent Educ. 2011 Nov;15 Suppl 1:23-31. doi: 10.1111/j.1600-0579.2011.00711.x. PMID 22023543